CLINICAL TRIAL: NCT00940264
Title: Laparoscopic Transvaginal Hybrid Cholecystectomy: a Prospective Data Collection.
Status: Completed | Type: Observational
Sponsor: Ignazio Tarantino (Other)
Responsible Party: Sponsor-Investigator, Ignazio Tarantino, M.D., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: EKSG08/060/2B
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Cholecystolithiasis; Cholecystitis
Keywords: symptomatic cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Given indication for cholecystectomy
  Interventions: Procedure: transvaginal hybrid cholecystectomy

INTERVENTIONS:
Procedure: transvaginal hybrid cholecystectomy — transvaginal hybrid cholecystectomy: using one trans-umbilical 5mm trocar and 2 (one 12mm trocar, one 5-mm trocar)inserted through the posterior colpotomy. Removal of the gallbladder through the transvaginal access.

SUMMARY:
Transvaginal hybrid procedures especially the transvaginal hybrid cholecystectomy are of interest as an available NOTES-Procedure for the clinical routine. Few authors have demonstrated the feasibility and safety in a selected patient collective. The aim of this prospective data collection is to evaluate the feasibility in the clinical routine in a non select patient collective.

Therefore all patients giving the informed consent to the transvaginal hybrid cholecystectomy will be included and assessed concerning feasibility to perform the transvaginal approach and complete the operation transvaginally.

ELIGIBILITY:
Inclusion Criteria:

* given informed consent for transvaginal hybrid cholecystectomy

Exclusion Criteria:

* pregnancy
* malignoma
* present choledocholithiasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patiens with given indication for cholcystectomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of the transvaginal operation | 30 days

SECONDARY OUTCOMES:
Long-term life quality and sexual dysfunction | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of surgery, Sankt Gallen, Switzerland